CLINICAL TRIAL: NCT06754475
Title: The Effect of Upper Extremity Low-Volume High-Intensity Interval Training on Physical and Cognitive Functions in Heart Failure Patients
Brief Title: Effects of Upper Extremity Low Volume HIIT in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nurel Ertürk, Assist. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/17
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: High Intensity Interval Training; Heart Failure; Exercises
Keywords: high intensity interval training; upper extremity; exercises capacity
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): İntervention Group: LV-HIIT
  Interventions: Other: Low-volume, high-intensity interval training
- Control group (Other): Control group
  Interventions: Drug: Standart medical treatment

INTERVENTIONS:
Other: Low-volume, high-intensity interval training — Low-volume, high-intensity interval training with an arm ergometer will be given two days a week for a total of eight weeks.
  Arms: Patients
Drug: Standart medical treatment — Standart medical teatment
  Arms: Control group

SUMMARY:
This study was planned to investigate the effects of upper extremity low-volume high-intensity interval training (LV-HIIT) on physical and cognitive function in patients with heart failure with preserved ejection fraction(HFpEF).The research was planned as a randomized controlled trial. Patients with clinically stable HFpEF at cardiology clinic will be included in the study. These cases will be randomly divided into two groups: intervention group and control grup. After 8 weeks intervention physical functions before and after treatment; functional exercise capacity, arm exercise capacities , peripheral muscle strength , fatigue cognitive functions; anxiety and depression and fear of movement will be evaluated.

DETAILED DESCRIPTION:
Patients in the DV-HIIT group will receive training consisting of 4 minutes of warm-up and cool-down at 50% Wmax on an arm ergometer, 1 minute of training at 85-95% Wmax work intensity, followed by 6 interval training periods including 1 minute of active recovery periods at 50-70% Wmax, 2 days/week, totaling 8 weeks of training. The control group will be followed with standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition stable for ≥4 weeks.
* New York Heart Association functional classification I-II to III
* Over 18 years old

Exclusion Criteria:

History of CABG surgery

* Unstable angina pectoris
* Severe arrhythmia
* Acute pericarditis, endocarditis, myocarditis
* Severe left ventricular failure (EF <40%)
* Acute pulmonary embolism
* History of syncope
* Dissecting aneurysm
* Thrombophlebitis
* Orthopedic disorders that may interfere with exercise
* Uncontrolled hypertension, severe pulmonary arterial hypertension
* Moderate-severe valve disease
* Decompensated Congestive Heart Failure
* Electrolyte abnormalities
* Hypertrophic Cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
maximal arm exercises capacity | At baseline and after 8 week
  maximal arm exercises capacity will measurement with arm ergometer test.
Functional capacity | At baseline and after 8 week
  Functional capacity will be assessed with the six-minute walk test (6MWT).
Upper extremity muscle strength | At baseline and after 8 week
  Upper extremity muscle strength will be evaluated with a digital dynamometer and hand grip strength will be evaluated with a jamar.
reaction time | At baseline and after 8 week
  The auditory and visual reaction times of the individuals will be determined. The instrument used during the test can give three stimuli and consists of two parts, In measuring the reaction times, care will be taken to ensure that the measurement area is a noiseless and light-receiving environment. Individuals will be told the technique of the test and will be asked to make 1 attempt against sound and light stimulation. After the trial, 3 measurements will be taken and the results will be recorded in milliseconds
cognitive function | At baseline and after 8 week
  Mini mental Questionaire will use. Min 24 point is the cut of for this test
Postural sway | At baseline and after 8 week
  The postural oscillations of the patients will be evaluated with the body oscillation device, which measures the oscillation in two axes. In this test, the participant will be asked to stand in the upright position with a distance of 10 cm between the two feet and to maintain your upright position for 30 seconds. The participant will be measured twice with the eyes open and closed. With these measurements, the mediolateral and anteroposterior oscillation distances of the patients will be measured and recorded on the computer
heart rate variablity | At baseline and after 8 week

SECONDARY OUTCOMES:
hand steadness | At baseline and after 8 week
  The auditory and visual reaction times of the individuals will be determined. The instrument used during the test can give three stimuli and consists of two parts, In measuring the reaction times, care will be taken to ensure that the measurement area is a noiseless and light-receiving environment. Individuals will be told the technique of the test and will be asked to make 1 attempt against sound and light stimulation. After the trial, 3 measurements will be taken and the results will be recorded in milliseconds.
Anxiety and depresion | At baseline and after 8 week
  Hospital anxiety and depression Scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). It is worth noting that items referring to depression symptoms that describe somatic aspects of depression (e.g. insomnia and weight loss) are not included in the scale.
activities of daily living | At baseline and after 8 week
  Nottingham Health Profile (NHP) will used. The questionnaire is divided into two parts. The first parts comprises 38 questions in six categories: sleep, physical mobility, energy, pain, emotional reactions, and social isolation.The second part of the NHP is made up of seven statements about areas of life that are commonly affected by health: paid employment, jobs around the house, social life, personal relationships, sex life, hobbies and interests, and holidays. Scores on the NHP can range from 0 i.e. no distress to 100 i.e severe distress.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Tarsus University, TARSUS, Mersin, Mersin, Mersin
  - Nurel Ertürk, TARSUS, Mersin, Yenişehir, Mersin

IPD SHARING:
Plan to Share IPD: No
All IPD collected throughout the trial, only IPD used in the results publication